CLINICAL TRIAL: NCT03707002
Title: Randomized, Placebo-controlled Double Blind Study to Evaluate the Effects of Dietary Supplementation With Short-chain Fructo-oligosaccharides (scFOS) on Nincrease in Stool Frequency in Constipated People
Brief Title: Effect of scFOS on Increase in Stool Frequency in Constipated People
Acronym: CONSYST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syral (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other); CreaBio Rhone-Alpes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PEC14513
Record Dates: First submitted 2018-10-05; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Functional Constipation; Healthy
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical sachets containing 5g of scFOS or placebo (maltodextrins)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scFOS (Active Comparator): scFOS consumed at 5g/day for 6 weeks
  Interventions: Dietary Supplement: scFOS
- Placebo (Placebo Comparator): maltodextrin consumed at 5g/day for 6 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: scFOS — daily intake for 6 weeks
  Arms: scFOS
Dietary Supplement: Maltodextrin — daily intake for 6 weeks
  Arms: Placebo

SUMMARY:
The study aims to evaluate the effects of short-chain fructo-oligosaccharides on the frequency and consistency of stools in subjects with functional constipation.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, double-blind study aims to evaluate the effects of short-chain fructo-oligosaccharides on the frequency and consistency of stools in subjects with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* functional constipation according to ROME III criteria with 3 or less than 3 stools per week
* BMI between 18 and 32kg/m², limits included
* Subjects who do not usually eat high-fibre foods
* Subjects who do not usually consume foods siad "reduced in sugars" or "light"
* Subjects who do not consume regularly pre- and probiotics in the form of dietary supplements

Exclusion Criteria:

* subjects presenting Irritable bowel syndrome
* history of chronic GI disorders: crohn disease, ulcerative colitis,....
* treatments likely to influence GI sensitivity or motility (laxative, neuroleptics,...)
* Antibiotic therapy in progress or in the past 8 weeks
* medical history with impact on the study objectives as defined by investigator
* known food allergy to one of the compounds of the study product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Stool frequency | 6 weeks
  Change in the number of stool per week between week at Baseline and the last week of supplementation

SECONDARY OUTCOMES:
Stool consistency | 6 weeks
  Change in the stool consistency between Baseline and the end of supplementation, (Bristol Stool Scale 1 = hard to 7 = watery)
Frequency and severity of Gastrointestinal symptoms | 6 weeks
  Change in the frequency (number of occurrence) and severity (Likert scores from 0= no symptom to 7 =severe symptoms) individual Gastro-Intestinal symptoms (bloating, abdominal pain, flatulence,...) between Baseline and the end of supplementation
Anxiety and depression | 6 weeks
  Changes in anxiety and depression score between Baseline and the end of supplementation, measured by HAD score (Zigmond et al, 1983, from 0 to 21, score above 11 = anxiety or depression related pathology

OTHER OUTCOMES:
Heart rate | at baseline and at the last visit (after 6 weeks)
  heart rate (bit per minute)
systolic blood pressure | at baseline and at the last visit (after 6 weeks)
  systolic blood pressure (mmHg)
diastolic blood pressure | at baseline and at the last visit (after 6 weeks)
  diastolic blood pressure (mmHg)
Adverse event | 6 weeks
  Registration of all adverse events (number and severity of events)

CONTACTS AND LOCATIONS:
Overall Officials: David Gendre, MD, Principal Investigator — BioFortis
Locations (1):
- Biofortis SAS, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No